CLINICAL TRIAL: NCT04387409
Title: A Phase III, Double-blind, Randomized, Placebo-controlled Multicentre Clinical Trial to Assess the Efficacy and Safety of VPM1002 in Reducing Healthcare Professionals' Absenteeism in the SARS-CoV-2 Pandemic by Modulating the Immune System
Brief Title: Study to Assess VPM1002 in Reducing Healthcare Professionals' Absenteeism in COVID-19 Pandemic
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Serum Life Science Europe GmbH (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VPM1002-DE-3.06CoV
Record Dates: First submitted 2020-05-11; First posted 2020-05-13 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Infection, Respiratory Tract
Keywords: infectious respiratory diseases; COVID-19
MeSH Terms: conditions — Respiratory Tract Infections; COVID-19 | interventions — VPM1002 recombinant BCG vaccine

STUDY DESIGN:
Intervention Model Description: Subjects who fulfil the inclusion/exclusion criteria will be centrally randomized in a 1:1 ratio to receive a single dose (0.1 ml) of either VPM1002 or Placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The reconstitution and administration of trial intervention will be done by unblinded site personnel who will not be involved in the collection or evaluation of outcome data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VPM1002 (Active Comparator): The active ingredient of the recombinant BCG vaccine, VPM1002, is Mycobacterium bovis rBCGΔureC::hly, freeze-dried and standardized to the number of viable mycobacteria (colony forming units; CFU) per application.
  Dose: 2-8 x 10e5 CFU VPM1002 administered in 0.1 ml reconstituted suspension.
  Interventions: Biological: VPM1002
- Placebo (Placebo Comparator): Physiological saline 0.1ml
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VPM1002 — The investigational product will be administered via intradermal injection with a 1.0-ml syringe, sub-graduated into hundredths of ml (1/100 ml), and fitted with a short bevel needle (25G/0.50 mm or 26G/0.45 mm, 10 mm in length).
  Arms: VPM1002
Biological: Placebo — The investigational product will be administered via intradermal injection with a 1.0-ml syringe, sub-graduated into hundredths of ml (1/100 ml), and fitted with a short bevel needle (25G/0.50 mm or 26G/0.45 mm, 10 mm in length).
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate whether vaccination of healthcare professionals with VPM1002 could reduce the number of days absent from work due to respiratory disease (with or without documented SARS-CoV-2 infection).

VPM1002 is a vaccine that is a further development of the old Bacillus Calmette-Guérin (BCG) vaccine, which has been used successfully as a vaccine against tuberculosis for about 100 years, especially in developing countries. VPM1002 has been shown in various clinical studies to be significantly safer than the BCG vaccine.

VPM1002 strengthens the body's immune defence and vaccination with BCG reduces the frequency of respiratory diseases. It is therefore assumed that a VPM1002 vaccination could also provide (partial) protection against COVID-19 disease caused by the new corona virus "SARS-CoV 2".

A total of 1200 health care professionals (doctors, nurses and paramedical staff) with high expected exposure to SARSCoV-2 infected patients will receive a single dose of either VPM1002 or Placebo. All subjects will be requested to enter data regarding absenteeism, adverse events / serious adverse events, hospitalizations, intensive care unit admissions into an online questionnaire.

DETAILED DESCRIPTION:
Based on the evidence that BCG vaccine

1. can potentiate immune responses to other vaccines through induction of trained innate immunity and heterologous adaptive immunity and
2. can reduce the incidence of respiratory infections, exert antiviral effects in experimental models, and reduce viremia in an experimental human model of viral infection,

it is hypothesized that BCG vaccination may induce (partial) protection against the susceptibility to and/or severity of SARS- CoV-2 infection.

VPM1002 is being developed with the aim to replace BCG by a vaccine that has a better safety profile and superior efficacy. Evidence from pre-clinical and clinical studies demonstrate that VPM1002 is safer and is more immunogenic than the existing BCG vaccine. It is therefore anticipated that VPM1002 will also perform better in reducing the severity of the symptoms of an infection with the SARS CoV-2 than the BCG vaccine. Further, manufacturing of VPM1002 using state-of-the-art production methods will help hasten the production of millions of doses in a very short time and thus would be beneficial in the current SARS-CoV-2 pandemic situation.

The current trial will assess the efficacy and safety of VPM1002 to reduce health care professionals ' absenteeism in the SARS-CoV-2 pandemic by modulating the immune system.

A total of 1200 health care professionals (doctors, nurses and paramedical staff) with high expected exposure to SARSCoV-2 infected patients (e.g. those employed in emergency departments, intensive care unit, infectious disease ward, COVID-19 isolation wards, respiratory wards, etc.) will be enrolled, across hospitals in Germany. Informed consent will be obtained from the subjects willing to take part in the trial. This will be followed by assessment of the eligibility criteria. Subjects who fulfil the inclusion/exclusion criteria will be centrally randomized in a 1:1 ratio to receive a single dose of either VPM1002 or Placebo.

All subjects will be requested to sign into a web-based tool designed for this trial. All subjects will be followed-up entirely remotely. The web-based questionnaires will be designed to collect data regarding absenteeism, adverse events / serious adverse events, hospitalizations, intensive care unit admissions and other secondary endpoints. The investigators will review the outcome and safety data.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* Male or female
* Hospital personnel with expected high SARS-CoV-2 exposure
* Subject is contractually capable, able to understand information on study and has signed informed consent sheet
* Subject has access to an internet-enabled electronic device
* Women of childbearing potential who are currently using reliable methods of birth control, have a negative pregnancy test during screening and have no intention to become pregnant for at least 3 months post-vaccination.

Exclusion Criteria:

* Known hypersensitivity or allergy to (components of) the VPM1002 vaccine or serious adverse reactions to prior BCG administration
* Known active or latent Mycobacterium tuberculosis infection or with another mycobacterial species. A history with or suspicion of M. tuberculosis infection.
* Fever (>38 °C) within the past 24 hours
* Pregnant or breast-feeding
* Suspicion of active viral or bacterial infection
* Participation of subject in another study within 30 days before screening and during this study
* Person is an employee of the sponsor, a relative of the investigator or in direct reporting line to clinical trial staff at the clinical trial site
* Severely immunocompromised subjects, such as:

  1. subjects with known infection with the human immunodeficiency virus (HIV);
  2. subjects with solid organ transplantation;
  3. subjects with bone marrow transplantation;
  4. subjects under chemotherapy, immunotherapy and radiotherapy;
  5. subjects with primary immunodeficiency;
  6. treatment with any anti-cytokine therapies;
  7. treatment with oral or intravenous steroids defined as daily doses of 10 mg prednisone or equivalent for longer than 3 months
* Active solid or non-solid malignancy or lymphoma in the past 5 years
* Direct involvement in the design or the execution of the present clinical trial
* Expected absence from work of ≥4 of the following 12 weeks due to any reason (holidays, maternity leave, retirement, planned surgery etc)
* Employed to the hospital < 22 hours per week
* Previous positive SARS-CoV-2 test result

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of days absent from work due to respiratory disease (with or without documented SARS-CoV-2 infection) | From day 0 to day 240

SECONDARY OUTCOMES:
Cumulative incidence of documented SARS-CoV-2 infection | From day 0 to day 240
Number of days absent from work due to documented SARS-CoV-2 infection | From day 0 to day 240
Number of days absent from work due to exposure to person with documented SARS-CoV-2 infection | From day 0 to day 240
Number of days absent from work due to symptoms of respiratory disease, documented SARS-CoV-2 infection, or fever (≥ 38 °C) | From day 0 to day 240
Number of days of self-reported fever (≥ 38 °C) | From day 0 to day 240
Number of days of self-reported acute respiratory symptoms | From day 0 to day 240
Cumulative incidence of self-reported acute respiratory symptoms | From day 0 to day 240
Cumulative incidence of death for any reason | From day 0 to day 240
Cumulative incidence of death due to documented SARS-CoV-2 infection | From day 0 to day 240
Cumulative incidence of ICU admission for any reason | From day 0 to day 240
Cumulative incidence of ICU admission due to documented SARS-CoV-2 infection | From day 0 to day 240
Cumulative incidence of hospital admission for any reason | From day 0 to day 240
Cumulative incidence of hospital admission due to documented SARS-CoV-2 infection | From day 0 to day 240

CONTACTS AND LOCATIONS:
Overall Officials: Leander Grode, Dr rer nat, Study Director — Serum Life Science Europe GmbH
Locations (3):
- Germany (3):
  - Ludwig-Maximilians-Universität München, München, Bavaria
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - SocraTec R&D GmbH, Erfurt, Thuringia

IPD SHARING:
Plan to Share IPD: No
There is uncertainty whether the European Union General Data Protection Regulation allows dissemination of individual participant data to other researchers. Some reasons why the EU Regulation would not allow this are the lack of suitable safeguards when person data are transferred to any researcher asking for it and the impairment of the rights of the subjects for erasure of their data once they are disseminated.